CLINICAL TRIAL: NCT01294397
Title: The Effects of Denosumab on the Pharmacokinetics of Etanercept in Postmenopausal Women With Low Bone Mineral Density and Rheumatoid Arthritis
Brief Title: Effects of Denosumab on the Pharmacokinetics of Etanercept
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of enrollment.
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20101324
Record Dates: First submitted 2011-01-13; First posted 2011-02-11 (Estimated); Results first posted 2017-06-20 (Actual); Last update posted 2017-06-20 (Actual); Status verified 2017-04

CONDITIONS: Postmenopausal; Osteopenia; Rheumatoid Arthritis; Osteoporosis
Keywords: Amgen; Phase 1; Postmenopausal; Osteopenia; Rheumatoid; Bone Mineral Density; Arthritis; Pharmacokinetics; Osteoporosis
MeSH Terms: conditions — Bone Diseases, Metabolic; Arthritis, Rheumatoid; Osteoporosis; Arthritis | interventions — Etanercept; Denosumab

ARMS (1):
- Etanercept + Denosumab (Experimental): Participants received etanercept 50 mg subcutaneously once weekly for 25 weeks. On study day 8, participants were administered a single 60 mg subcutaneous injection of denosumab.
  Interventions: Drug: Etanercept; Drug: Denosumab

INTERVENTIONS:
Drug: Etanercept — Administered by subcutaneous injection once a week
  Other Names: Enbrel®
Drug: Denosumab — Administered by subcutaneous injection
  Other Names: Prolia®

SUMMARY:
The primary objective of the study was to characterize the effects of a single dose of denosumab on the pharmacokinetics (PK) of etanercept in postmenopausal women with low bone mineral density (BMD) and rheumatoid arthritis based on area under the serum concentration-time curve (AUC) and maximum observed serum concentration (Cmax).

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women (postmenopausal is defined as no vaginal bleeding or spotting for at least 12 months)
* Low bone mineral density (BMD) as determined by screening BMD T-scores of the lumbar spine (L1 to L4), or total evaluable vertebrae (if fewer than L1 to L4), or total hip ≤ -1.0
* Receiving a 50 mg dose of etanercept once weekly ≥ 6 months prior to screening and expected to continue etanercept treatment at this dose and frequency through end of study (EOS)
* If currently taking methotrexate (MTX), receiving a stable dose (7.5 to 20 mg/week) of MTX ≥ 8 weeks prior to screening
* Willing and able to take ≥ 1,000 mg elemental calcium and ≥ 400 IU vitamin D daily upon enrollment

Exclusion Criteria:

* Type 1 diabetes; OR poorly controlled Type 2 diabetes (hemoglobin A1c (HbA1c) > 8.0% at screening; HbA1c ≤ 8.0% within 6 months of screening is acceptable if supporting laboratory documentation is available)
* History of heart failure, coronary artery bypass graft, or cardiac arrhythmia; OR history of acute coronary syndrome
* Comorbid autoimmune disease, demyelinating disease, or hematologic abnormalities
* History of joint replacement in hand and/or wrist; OR history of fused joint in hand and/or wrist
* Prior history or current evidence of osteonecrosis/osteomyelitis of the jaw; OR active dental or jaw condition that requires oral surgery, or non-healed dental/oral surgery; OR planned invasive dental procedure(s) during the course of the study
* Previous exposure to denosumab

Ages: 45 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-03; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (2):
- United States (2):
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Dallas, Texas

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 2 centers in the United States. The first participant enrolled on 07 March 2011; the last participant was enrolled on 15 June 2015.
Pre-assignment Details: Following determination of eligibility at screening, 19 participants were enrolled into a 4-week run-in period of etanercept 50 mg subcutaneous once-weekly injection to ensure steady-state.
Period: Overall Study
Arm/Group | Etanercept + Denosumab
Started | 19
Completed | 17
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Administrative Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Etanercept + Denosumab
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic/Latino | 1
  Not Hispanic/Latino | 18
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Black (or African American) | 1
  Mixed race | 0
  Native Hawaiian or Other Pacific Islander | 0
  White | 18

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Serum Concentration-time Curve From 0 to 168 Hours (AUC0-168) for Etanercept
Description: The AUC0-168 of etanercept was measured when administered alone (assessed from day 1) and after administration with denosumab (assessed from day 22, 14 days after denosumab dosing, close to the time of the maximum observed denosumab serum concentration and corresponding to a time approximately 1 week after maximal pharmacodynamic (PD) effects of denosumab are attained).
Time Frame: Day 1 and day 22; at each time point samples were taken predose and 2, 3, 4, 5, 6 and 8 days postdose.
Population: Participants with available AUC data
Measure: Mean (Standard Deviation); unit: day*μg/mL
Arm/Group | Etanercept + Denosumab
Number analyzed (Participants) | 17
day*μg/mL
  Etanercept Alone (Day 1) | 40.8 (18.8)
  Etanercept + Denosumab (Day 22) | 40.4 (26.6)
Statistical Analysis 1: Comparison: Etanercept + Denosumab; Log-transformed AUC0-168 was analyzed with a mixed-effects model with treatment as the fixed effect and subject as the random effect. The mean difference between day 22 and day 1 was expressed as a percentage of the reference (day 1). The mean differences and the 90% CIs were back transformed to produce the ratio (day 22 vs. day 1) of the geometric means and the 90% CIs. If the CI for the ratio was within the standard acceptance range of 0.80 to 1.25, absence of an interaction was concluded; Test type: Superiority or Other; Least Squares Mean Ratio of Day 22/Day 1 = 0.96, 90% CI 2-sided [0.85 to 1.08] — Two one-sided tests

2. Primary Outcome: Maximum Observed Serum Concentration (Cmax) of Etanercept
Time Frame: Day 1 and day 22; at each time point samples were taken predose and 2, 3, 4, 5, 6 and 8 days postdose.
Population: Participants with available Cmax data
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Etanercept + Denosumab
Number analyzed (Participants) | 19
μg/mL
  Etanercept Alone - Day 1 (n=19) | 8.71 (5.47)
  Etanercept + Denosumab - Day 22 (n=18) | 8.25 (5.57)
Statistical Analysis 1: Comparison: Etanercept + Denosumab; Log-transformed Cmax was analyzed with a mixed-effects model with treatment as the fixed effect and subject as the random effect. The mean difference between day 22 and day 1 was expressed as a percentage of the reference (day 1). The mean differences and the 90% CIs were back transformed to produce the ratio (day 22 vs. day 1) of the geometric means and the 90% CIs. If the CI for the ratio was within the standard acceptance range of 0.80 to 1.25, absence of an interaction was concluded; Test type: Superiority or Other; Least Squares Mean Ratio of Day 22/Day 1 = 0.92, 90% CI 2-sided [0.81 to 1.05] — Two one-sided tests

3. Secondary Outcome: Time to Maximum Serum Concentration (Tmax) of Etanercept
Time Frame: Day 1 and day 22; at each time point samples were taken predose and 2, 3, 4, 5, 6 and 8 days postdose.
Population: Participants with available Tmax data
Measure: Median (Full Range); unit: days
Arm/Group | Etanercept + Denosumab
Number analyzed (Participants) | 19
days
  Etanercept Alone - Day 1 (n=19) | 3.0 [0.99 to 4.9]
  Etanercept + Denosumab - Day 22 (n=18) | 2.0 [0.93 to 4.9]

4. Secondary Outcome: Serum Denosumab Concentration
Time Frame: Prior to etanercept and denosumab dose administrations, as applicable, on days 8, 22, and 29
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Etanercept + Denosumab
Number analyzed (Participants) | 19
μg/mL
  Day 8 (n=19) | 0.00 (0.00)
  Day 22 (n=18) | 5.30 (1.35)
  Day 29 (n=18) | 4.85 (1.35)

5. Secondary Outcome: Percent Change From Baseline in Serum C-telopeptide (sCTx) Concentrations
Time Frame: Baseline (Day 8) and Days 22, 29, 85, and 176
Population: Participants with available data at baseline (19) and each time point (indicated by n)
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Etanercept + Denosumab
Number analyzed (Participants) | 19
percent change
  Day 22 (n = 18) | -32.3 [-58.7 to 0.0]
  Day 29 (n = 18) | -32.3 [-60.9 to 0.0]
  Day 85 (n = 17) | -26.2 [-60.9 to 0.0]
  Day 176/End of Study (n = 19) | -25.1 [-60.4 to 0.0]

ADVERSE EVENTS:
Time Frame: From first dose of etenercept in the run-in period (day -28) until end of study (day 176).
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- Etanercept 50 mg Day - 28 - Day 7: Participants received etanercept 50 mg subcutaneously once weekly. Adverse events are reported from day -28 until day 7.
- Etanercept 50 mg + Denosumab 60 mg Day 8 - EOS: Participants received etanercept 50 mg subcutaneously once weekly. On study day 8, participants were administered a single 60 mg subcutaneous injection of denosumab.
  Adverse events are reported from day 8 to end of study (day 176).
- All Subjects On-study: Participants received etanercept 50 mg subcutaneously once weekly for 25 weeks. On study day 8, participants were administered a single 60 mg subcutaneous injection of denosumab.
  Adverse events are reported from day -28 up to day 176.
Arm/Group | Etanercept 50 mg Day - 28 - Day 7 | Etanercept 50 mg + Denosumab 60 mg Day 8 - EOS | All Subjects On-study
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 13/19 | 2/19 | 13/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept 50 mg Day - 28 - Day 7 (N=19) | Etanercept 50 mg + Denosumab 60 mg Day 8 - EOS (N=19) | All Subjects On-study (N=19)
Eye haemorrhage (Eye disorders) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Injection site erythema (General disorders) | 1 | 0 | 1
Injection site pruritus (General disorders) | 1 | 0 | 1
Nodule (General disorders) | 1 | 0 | 1
Seasonal allergy (Immune system disorders) | 1 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 1
Conjunctivitis (Infections and infestations) | 1 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 0 | 3
Urinary tract infection (Infections and infestations) | 2 | 0 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 1 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Fracture treatment (Surgical and medical procedures) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.